CLINICAL TRIAL: NCT07151456
Title: Short-term vs Conventional Glucocorticoid Therapy for the Treatment of the Initial Episode of Adult Patient With Steroid-sensitive Idiopathic Nephrotic Syndrome
Brief Title: Short-term gluCOCOrticoid in Adult STEROID-sensitive Nephrotic Syndrome: The COCO-ASTEROID Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Tianxin Chen, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-303
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Nephrotic Syndrome
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional course prednisolone arm (Active Comparator)
  Interventions: Drug: Conventional 24-week glucocorticoid regimen
- short-term course prednisolone arm (Experimental)
  Interventions: Drug: short-term course (12 week) glucocorticoid regimen

INTERVENTIONS:
Drug: Conventional 24-week glucocorticoid regimen — Weeks 1 - 4, Prednisolone 1mg/kg/day (max 80mg); Weeks 5 - 6: Prednisolone 0.8mg/kg/day (max 60mg); Weeks 7 - 8: Prednisolone 0.6mg/kg/day (max 50mg); Weeks 9 - 10: Prednisolone 0.5mg/kg/day (max 40mg); Weeks 11 - 12: Prednisolone 0.4mg/kg/day (max 30mg); Weeks 13 - 16: Prednisolone 0.3mg/kg/day (max 25mg); Weeks 17 - 20: Prednisolone 0.2mg/kg/day (max 15 Weeks 21 - 24: Prednisolone 0.1mg/kg/day (max 10mg).
  Arms: conventional course prednisolone arm
Drug: short-term course (12 week) glucocorticoid regimen — Weeks 1 - 4, Prednisolone 1mg/kg/day (max 80mg); Weeks 5-8: Prednisolone 1mg/kg/day (max 80mg) on alternate days; 9-12: Prednisolone 0.5mg/kg/day (max 40mg) on alternate days
  Arms: short-term course prednisolone arm

SUMMARY:
This study will compare a short-term course (12 week) glucocorticoid regimen with the Conventional 24-week regimen as originally proposed by KDIGO. The purpose of the study is to determine a short-term course (12 week) of glucocorticoid decreases the time to first relapse in adults presenting with steroid sensitive nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Urine protein: creatinine ratio ≥3000mg/g (300mg/mmol)
* Serum/plasma albumin level < 30g/L
* Age ≥ 16 years at the time of diagnosis
* No prior therapy with steroids, immunosuppressive or cytotoxic agents for any form of renal disease (other than the 28 days of prednisolone therapy given initially as routine clinical practice)
* No evidence of underlying systemic disorder or exposure to agents known to be associated with newly presenting steroid sensitive nephrotic syndrome
* Informed consent
* SSNS defined as Complete remission within 4 weeks of prednisone or prednisolone at standard dose

Exclusion Criteria:

* Secondary nephrotic syndrome
* Contradictions for glucocorticoids
* SRNS: Lack of complete remission within 4 weeks of therapy with daily prednisone or prednisolone at standard dose
* anti-PLA2R positive
* Adults with histological changes other than minimal lesion or focal segmental glomerular sclerosis (FSGS) glomerulonephritis where renal biopsy has been undertaken
* Adults with a prior history of poor compliance with medical therapy Known allergy to glucocorticoid therapy
* Other situations where the researcher deems it inappropriate to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Relapse | through study completion, an average of 2 years
  Relapse of proteinuria is defined by Albustix positive proteinuria (+++ or greater) for 3 consecutive days or the presence of generalised oedema plus 3+ proteinuria.

SECONDARY OUTCOMES:
Relapse rate | 12 months，24 months
  the proportion of adults who develop relapsing

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans JHC, Long E. A national audit of nephrotic syndrome: The initial course of prednisolone and outcome. Abstract. Ped Nephrol 1998;12(7):C154
- [Background] Hodson EM, Knight JF, Willis NS, Craig JC. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2004;(2):CD001533. doi: 10.1002/14651858.CD001533.pub2. PMID 15106158
- [Background] Ksiazek J, Wyszynska T. Short versus long initial prednisone treatment in steroid-sensitive nephrotic syndrome in children. Acta Paediatr. 1995 Aug;84(8):889-93. doi: 10.1111/j.1651-2227.1995.tb13787.x. PMID 7488812
- [Background] Bargman JM. Management of minimal lesion glomerulonephritis: evidence-based recommendations. Kidney Int Suppl. 1999 Jun;70:S3-16. doi: 10.1046/j.1523-1755.1999.07002.x. PMID 10369190
- [Background] Abramowicz M, Barnett HL, Edelmann CM Jr, Greifer I, Kobayashi O, Arneil GC, Barron BA, Gordillo-P G, Hallman N, Tiddens HA. Controlled trial of azathioprine in children with nephrotic syndrome. A report for the international study of kidney disease in children. Lancet. 1970 May 9;1(7654):959-61. doi: 10.1016/s0140-6736(70)91093-7. No abstract available. PMID 4191931
- [Background] Brodehl J. Conventional therapy for idiopathic nephrotic syndrome in children. Clin Nephrol. 1991;35 Suppl 1:S8-15. PMID 1860269
- [Background] Consensus statement on management and audit potential for steroid responsive nephrotic syndrome. Report of a Workshop by the British Association for Paediatric Nephrology and Research Unit, Royal College of Physicians. Arch Dis Child. 1994 Feb;70(2):151-7. doi: 10.1136/adc.70.2.151. No abstract available. PMID 8129444
- [Background] Trompeter RS, Lloyd BW, Hicks J, White RH, Cameron JS. Long-term outcome for children with minimal-change nephrotic syndrome. Lancet. 1985 Feb 16;1(8425):368-70. doi: 10.1016/s0140-6736(85)91387-x. PMID 2857421